CLINICAL TRIAL: NCT00923806
Title: Phase I/II Study of Metastatic Cancer That Expresses Carcinoembryonic Antigen (CEA) Using Lymphodepleting Conditioning Followed by Infusion of Anti-CEA TCR-Gene Engineered Lymphocytes
Brief Title: Gene Therapy Using Anti-CEA Cells to Treat Metastatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to poor accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090047; 09-C-0047; NCT00809978 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Cancer
Keywords: Metastatic Cancer; Tumor Regression; Safety; Immunotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gene Therapy Treatment (Experimental)
  Interventions: Biological: PG13-CEA_TCR (Anti-CEA TCR PBL); Drug: Aldesleukin

INTERVENTIONS:
Biological: PG13-CEA_TCR (Anti-CEA TCR PBL)
Drug: Aldesleukin — 720,000 IU/kg intravenous over 15 minutes every 8 hours for up to 5 days
  Other Names: Proleukin

SUMMARY:
Background:

* Carcinoembryonic antigen (CEA) is a protein present mostly in cancer cells.
* An experimental procedure developed for treating patients with cancer uses blood cells found in their tumors or bloodstream. These cells are genetically modified using the anti-CEA gene and a type of virus. The modified cells (anti-CEA cells) are grown in the laboratory and then given back to the patient to try to decrease the size of the tumors. This is called gene therapy.

Objectives:

* To determine whether advanced cancers that that express the CEA antigen can be treated effectively with lymphocytes (white blood cells) that have been genetically engineered to contain an anti-CEA protein.

Eligibility:

* Patients 18 years of age and older with metastatic cancer (cancer that has spread beyond the original site) and for whom standard treatments are not effective.
* Patients' tumors express the CEA antigen.
* Patients have the human leukocyte (HLA-A*0201) antigen.

Design:

* Workup with scans, x-rays and other tests.
* Leukapheresis to obtain cells for preparing the anti-CEA cells for later infusion.
* 1 week of chemotherapy to prepare the immune system for receiving the anti-CEA cells.
* Infusion of anti-CEA cells, followed by interleukin-2 (IL-2) treatment. The cells are given as an infusion through a vein. IL-2 is given as a 15-minute infusion through a vein every 8 hours for a maximum of 15 doses.
* 1-2 weeks of recovery from the effects of chemotherapy and IL-2.
* Periodic follow-up clinic visits after hospital discharge for physical examination, review of treatment side effects, laboratory tests and scans every 1 to 6 months.

DETAILED DESCRIPTION:
Background:

* We have constructed a single retroviral vector that contains both the alpha and beta chains of a T cell receptor (TCR) that recognizes the carcinoembryonic antigen (CEA), which can be used to mediate genetic transfer of this TCR with high efficiency (greater than 30%) without the need to perform any selection.
* In co-cultures with HLA-A2 and CEA positive tumors, anti-CEA TCR transduced T cells secreted significant amounts of interferon-gamma (IFN-gamma) with high specificity.

Objectives:

Primary objectives:

* To evaluate the safety of the administration of anti-CEA TCR engineered peripheral blood lymphocytes in patients receiving the non-myeloablative conditioning regimen and aldesleukin.
* To determine if the administration of anti-CEA TCR engineered peripheral blood lymphocytes and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer that expresses CEA.
* To determine the in vivo survival of TCR gene-engineered cells.

Secondary objective:

- To determine the in vivo survival of TCR gene-engineered cells.

Eligibility:

Patients who are HLA-A*0201 positive and 18 years of age or older must have

* metastatic cancer whose tumors express the CEA antigen where the life limiting component of the disease is hepatic metastases;
* previously received and have been a non-responder to or recurred to standard care for metastatic disease;

Patients should not have:

- contraindications for high dose aldesleukin administration.

Design:

* Peripheral blood mononuclear cells (PBMC) obtained by leukapheresis (approximately 5 times 10(9) cells) will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of approximately 10(8) to 5 times 10(8) cells to retroviral vector supernatant containing the anti-CEA TCR genes.
* Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous (IV) infusion of ex vivo tumor reactive, TCR gene-transduced PBMC plus IV aldesleukin (720,000 IU/kg q8h for a maximum of 15 doses). Patients will receive CD8-enhanced anti-CEA TCR transduced cells.
* Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment. If the patient has stable disease (SD) or tumor shrinkage, repeat complete evaluations will be performed every 1-3 months. After the first year, patients continuing to respond will continue to be followed with this evaluation every 3-4 months until off study criteria are met.
* The study will be conducted using a Phase I/II optimal design. The protocol will proceed in a phase 1 dose escalation design, with six cohorts. Should a single patient experience a dose limiting toxicity (DLT) at a particular dose level, three more patients would be treated at that 3 dose to confirm that no greater than 1/6 patients have a DLT prior to proceeding to the next higher level. If a level with 2 or more DLTs in 3-6 patients has been identified, three additional patients will be accrued at the next-lowest dose, for a total of 6, in order to further characterize the safety of the maximum tolerated dose (MTD) prior to starting the phase II portion. If a DLT occurs in the first cohort, that cohort will be expanded to 6 patients. If 2 DLTs are encountered in this cohort, patients will be accrued to the de-escalation cohort.
* Once the MTD has been determined, the study then would proceed to the phase II portion. Patients will be entered into two cohorts based on histology: cohort 1 will include patients with metastatic colorectal cancer, and cohort 2 will include patients with other types of metastatic cancer that express CEA.
* For each of the 2 strata evaluated, the study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. For each of these two arms of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.
* The objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, and anti-CEA TCR-gene engineered lymphocytes is able to be associated with a clinical response rate that can rule out 5% (p0=0.05) in favor of a modest 20% partial response (PR) + complete response (CR) rate (p1=0.20).

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Metastatic cancer that expresses carcinoembryonic antigen (CEA) as assessed by one of the following methods:

   * Immunohistochemistry of resected tissue, assessed by immunohistochemistry (IHC) in the Clinical Laboratory Improvement Amendments (CLIA) approved test in the Laboratory of Pathology, Center for Cancer Research (CCR), National Cancer Institute (NCI), National Institutes of Health (NIH). Since the affinity of the antibody is weak, a result of greater than or equal to 1+ is considered positive.
   * Detection of elevated levels of circulating CEA using a standard clinical enzyme-linked immunosorbent (ELISA) assay. Results will be considered positive if CEA level is greater than 10 mcg/L.
   * Metastatic cancer diagnosis will be confirmed by the Laboratory of Pathology at the NCI.
2. Hepatic metastases must represent the life limiting components of the disease defined as liver disease with a very high likelihood of causing the death of a patient according to the best clinical judgment of the attending physician.
3. Patients must have previously received systemic standard care (or effective salvage chemotherapy regimens) for metastatic disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred.
4. Greater than or equal to 18 years of age.
5. Willing to sign a durable power of attorney
6. Able to understand and sign the Informed Consent Document
7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
8. Life expectancy of greater than three months.
9. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the preparative regimen.
10. Patients must be human leukocyte antigen (HLA-A*0201) positive
11. Serology:

    1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    2. Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.
12. Hematology:

    1. Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
    2. White blood cell (WBC) (greater than 3000/mm^3.
    3. Platelet count greater than 100,000/mm^3.
    4. Hemoglobin greater than 8.0 g/dl.
13. Chemistry:

    1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
    2. Serum creatinine less than or equal to 1.6 mg/dl.
    3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
14. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
2. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent systemic steroid therapy
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of coronary revascularization or ischemic symptoms
8. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.
9. Documented LVEF of less than or equal to 45% tested in patients with:

   1. History of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
   2. Age greater than or equal to 60 years old
10. Documented forced expiratory volume (FEV1) less than or equal to 60% predicted tested in patients with:

    1. A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
    2. Symptoms of respiratory dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
clinical response of the administration of anti-CEA TCR engineered peripheral blood lymphocytes in patients receiving the non-myeloablative conditioning regimen and aldesleukin in patients with metastatic cancer.

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dudley ME, Wunderlich JR, Robbins PF, Yang JC, Hwu P, Schwartzentruber DJ, Topalian SL, Sherry R, Restifo NP, Hubicki AM, Robinson MR, Raffeld M, Duray P, Seipp CA, Rogers-Freezer L, Morton KE, Mavroukakis SA, White DE, Rosenberg SA. Cancer regression and autoimmunity in patients after clonal repopulation with antitumor lymphocytes. Science. 2002 Oct 25;298(5594):850-4. doi: 10.1126/science.1076514. Epub 2002 Sep 19. PMID 12242449
- [Background] Gattinoni L, Powell DJ Jr, Rosenberg SA, Restifo NP. Adoptive immunotherapy for cancer: building on success. Nat Rev Immunol. 2006 May;6(5):383-93. doi: 10.1038/nri1842. PMID 16622476
- [Background] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326